CLINICAL TRIAL: NCT05072431
Title: Examining the Effectiveness of 3D Virtual Reality Training on Problem-solving, Self-efficacy, and Teamwork Among Inexperienced Volunteers Helping With Drug Use Prevention: Randomized Controlled Trial
Brief Title: The Effectiveness of 3D VR Training System for Supporting Volunteers on Adolescents' Illegal Drug Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201805HS007
Record Dates: First submitted 2021-09-28; First posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-09

CONDITIONS: Illicit Drugs
Keywords: 3D virtual reality; Supporting volunteers; Problem solving; Self-efficacy; Teamwork
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The participants in the experimental group received the 3D VR training program.
  Interventions: Other: SVVR training program
- Control group (No Intervention): The control group did not receive any intervention.

INTERVENTIONS:
Other: SVVR training program — The SVVR training program is consisted of five scenarios with tasks. Before the SVVR training implementation, the research team provided 10-minute orientation session to introduce the purpose of the training. The 3D VR professional taught the participants how to wear the 3D VR helmets and select the VR scenes, so that the participants could practice multiple times.
  Arms: Experimental group

SUMMARY:
The purpose of that study was to apply the 3D virtual reality technology to develop a training program aiming at improving the abilities of problem solving, self-efficacy and teamwork of supervisory volunteers on adolescents' illegal drug use.

DETAILED DESCRIPTION:
Use of illegal drug among adolescents is one of the critical health problems in this age group. The purpose of that study was to apply the 3D virtual reality technology to develop a training program aiming at improving the abilities of problem solving, self-efficacy and teamwork of supervisory volunteers on adolescents' illegal drug use. This study used a randomized controlled design with recruiting 68 participants. The participants in the experimental group received the 3D VR training program and the counterparts in the control group did not receive any intervention. The participants in the experimental group performed better on problem solving, self-efficacy and teamwork. In addition, the scores of technology use related variables also supported that experimental participants favored the 3D VR training system. The findings suggested that the 3D VR training system enhanced the supporting volunteers' abilities to deal with adolescents' illegal drug use. The 3D VR program showed potential for future promotion to supporting volunteers that contribute to improve volunteers' abilities on dealing with adolescents' illegal drug use.

ELIGIBILITY:
Inclusion Criteria:

* accompanies at least an adolescent with drug use to
* having less than 2 year of supporting experiences
* having experiences of using technology products
* able to operate SVVR.

Exclusion Criteria:

* the volunteers who were suffering from cybersickness.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
The task characteristics | about one month
  Referenced related literatures (Goodhue, 1995) (Goodhue, 1995), developed 「The task technology characteristics」scale, a total of 3 questions, the task technology characteristics mainly understand the participants' experience in drug use students and related training, the higher scores indicated that participants are experienced in drug use students and related training.
Problem-solving skills | about one month
  Referenced relevant literatures (Association of American Colleges & Universities, 2009)(Association of American Colleges & Universities, 2009), developed「Problem-solving skills」scale, a total of 6 questions, The problem-solving skills mainly understand the participants' problem-solving skills in drug use students , the higher scores indicated that participants have better abilities.
Self-efficacy | about one month
  Referenced related literatures (Schwarzer, Bäßler, Kwiatek, Schröder, & Zhang, 1997)(Schwarzer, Bäẞler, Kwiatek, Schröder, & Zhang,1997), developed「Self-efficacy」scale, a total of 6 questions, The Self-efficacy mainly understand the participants' confidence in counseling drug use students, the higher scores demonstrated the more confident participants were
Team cooperation | about one month
  Referenced relevant literatures (Hughes & Jones, 2011)(Hughes & Jones, 2011), developed「Team cooperation」scale, a total of 4 questions, The Team cooperation mainly understand the participants' Team cooperation abilities in drug use students , the higher scores indicated that participants have better Team cooperation abilities.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chiang CH, Huang CM, Sheu JJ, Liao JY, Hsu HP, Wang SW, Guo JL. Examining the Effectiveness of 3D Virtual Reality Training on Problem-solving, Self-efficacy, and Teamwork Among Inexperienced Volunteers Helping With Drug Use Prevention: Randomized Controlled Trial. J Med Internet Res. 2021 Nov 2;23(11):e29862. doi: 10.2196/29862. PMID 34726606